CLINICAL TRIAL: NCT05330988
Title: Effects of tDCS on Post-stroke Fatigue and Inflammation
Brief Title: Post-stroke Fatigue, Inflammation, tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center of Neuromodulation for Rehabilitation (Other)
Responsible Party: Principal Investigator, John H Kindred, Principle Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00118687; P2CHD086844 (NIH)
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Fatigue; Chronic Stroke; Stroke Sequelae
MeSH Terms: conditions — Stroke; Fatigue | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Real (Experimental): Randomly selected participants will receive 20 min. of anodal transcranial direct current stimulation to the the top of their heads. The current will slowly be ramped up over 30 secs.
  Interventions: Device: anodal transcranial direct current stimulation (a-tDCS)
- Sham (Sham Comparator): Randomly selected participants will receive 20 min. of sham transcranial direct current stimulation to the top of their heads. Sham stimulation is accomplished by turning on the device and slowly increasing and subsequently decreasing the amount of current to zero. This occurs over 30 secs.
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: anodal transcranial direct current stimulation (a-tDCS) — The 1x1 platform is the most state-of-the-art, customizable, and reliable platform for pad-based Transcranial Electrical Stimulation.
  Other Names: 1x1 - tDCS, Soterix Medical, US Patents: US9956395B2, US8818515B2, US8718778B2.
  Arms: Real
Device: sham stimulation — The 1x1 platform is the most state-of-the-art, customizable, and reliable platform for pad-based Transcranial Electrical Stimulation.
  Other Names: 1x1 - tDCS, Soterix Medical, US Patents: US9956395B2, US8818515B2, US8718778B2.
  Arms: Sham

SUMMARY:
Fatigue is a common condition after an individual has a stroke. While the negative impacts of post-stroke fatigue are well known, the knowledge of the causes of post-stroke fatigue and effective treatments for post-stroke fatigue are lacking. This small study will investigate the possible benefits of transcranial direct current stimulation (tDCS), which uses small electrical currents supplied by a 9-volt battery, on post-stroke fatigue and investigate tDCS' possible anti-inflammatory effects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of any race or ethnicity
* 35-80 years of age
* 6+ months post-stroke
* Have clinically present fatigue for 6 months
* Able to walk 10m unassisted

Exclusion Criteria:

* Absolute contraindications to MRI, TMS (transcranial magnetic stimulation), or tDCS (e.g., implanted metal devices, history of seizure, and surgical clips or staples)
* Inability to understand and provide written informed consent
* Multiple strokes on opposite hemispheres
* Diagnosed comorbid neurological conditions (e.g. multiple sclerosis, Parkinson's disease, and dementia)
* Severe hypertension
* Cerebellar or brainstem strokes/lesions
* Concurrent depression and/or anxiety disorders

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Kindred, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that underlie the results reported in the article, after de-identification.
Supporting Information: Study Protocol, CSR
Time Frame: Immediately following publication no end date
Access Criteria: anyone who wishes to access the data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real | Sham
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real | Sham | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (6) | 63 (12) | 62 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Fatigue Severity Scale (FSS) Score
Description: Patient reported outcome measuring trait fatigue over the past 7 days. Minimum score = 7 maximum score = 63, higher scores indicate greater fatigue
Time Frame: Baseline, post-intervention (2-weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real | Sham
Number analyzed (Participants) | 6 | 6
units on a scale | -0.4 (0.9) | 0.2 (0.4)

2. Secondary Outcome: Change in Fatigue Assessment Scale (FAS)
Description: Patient reported outcome measuring trait fatigue. Minimum score = 10 maximum score = 50, higher scores indicate greater fatigue
Time Frame: Baseline, post-intervention (2-weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real | Sham
Number analyzed (Participants) | 6 | 6
score on a scale | -7 (8) | -4 (10)

ADVERSE EVENTS:
Time Frame: AEs were recorded before and immediately after each treatment session (5 days) by research staff administering the treatment. During follow-up, AEs were recorded during phone calls at 7, 14, and 28 days after an individual's last treatment session.
Arm/Group | Real | Sham
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT05330988/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT05330988/ICF_000.pdf